CLINICAL TRIAL: NCT06423053
Title: A Randomized Controlled Trial of a College Human Physiology Course With Integrated Mindfulness Practice on Student Applied Mindfulness and Stress Regulation (2025)
Brief Title: Mindfulness in a College Physiology Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Diane Gilbert-Diamond, Professor, Principal Investigator, Trustees of Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00032944
Record Dates: First submitted 2024-03-21; First posted 2024-05-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mindfulness; Stress; Perceived Stress; College Student Mental Health
Keywords: Mindfulness; College student; Stress; Applied mindfulness

STUDY DESIGN:
Intervention Model Description: The intervention group will consist of students enrolled in the Mindful Physiology course (Biology 3) at Dartmouth College in the spring 2025 term (3/31/2025- 6/4/2025). The control group will enroll students waitlisted for the course during the Spring 2025 term. The control participants will receive university wellness resources as usual. These include access to counseling and psychotherapy services at the university's counseling center, wellness advising at the student wellness center, and campus-wide wellness programs, such as weekly group yoga and meditation sessions and a free subscription to the Headspace app.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biology 3 students (Experimental): This arm consists of students enrolled in the Mindful Physiology course (Biology 3) at Dartmouth College during the Spring 2025 term who will have access to the course offerings and usual university wellness resources.
  Interventions: Behavioral: Biology Course with Integrated Mindfulness
- Biology 3 waitlisted students (No Intervention): This arm consists of students waitlisted for the Biology 3 course during the Spring 2025 term. They will receive university wellness resources as usual. These include access to wellness counselors, mental health advisors, and psychiatrists at the university's counseling center, wellness advising at the student wellness center, and campus-wide wellness programs, such as weekly group yoga and meditation sessions and a free subscription to the Headspace app. On-campus mindfulness retreats will also be advertised and accessible to the control group.

INTERVENTIONS:
Behavioral: Biology Course with Integrated Mindfulness — The intervention, Mindful Physiology, is an undergraduate-level biology course embedded with mindfulness practices. There will be 19 class sessions, each 1 hour and 50 minutes long, over 10 weeks. Students will be taught human physiology through didactic lectures, laboratory activities, and written quizzes typical for a college course. Each class meeting will have ~20 minutes of mindfulness practice in Thích Nhất Hạnh's Plum Village tradition. Students will also be encouraged to practice mindfulness for 15 minutes daily outside the class. Students will complete a daily log of their mindfulness practice and be given credit for each log completion regardless of the minutes of mindfulness practice. Students will be assigned a weekly written reflection on the physiology course content and/or their mindfulness practice. All students in the class are required to attend a 4.5-hour or a two-day (16-hour) on-campus mindfulness retreat.
  Arms: Biology 3 students

SUMMARY:
This proposed study aims to evaluate whether integrating mindfulness into an undergraduate biology course (Mindful Physiology) influences student applied mindfulness and stress regulation.

The primary questions are

1. Would completing the Mindful Physiology course increase applied mindfulness?
2. Would completing the course increase self-efficacy in stress regulation?
3. Would completing the course reduce perceived reactivity to acute stressors?

DETAILED DESCRIPTION:
The proposed study aims to evaluate whether integrating mindfulness practice into an undergraduate biology course influences student levels of applied mindfulness and stress regulation self-efficacy. A two-arm design will look at students who receive the intervention (a 10-week biology course with integrated mindfulness practice) and a control group of waitlisted students for the course who will only receive university wellness resources. Participants all attempted to register for the course during a set course selection period at the college and were randomly registered or waitlisted by the College Registrar. Students registered and waitlisted for the course will be recruited for the study, and those who provide informed consent will be enrolled. Data on applied mindfulness and stress regulation self-efficacy will be collected at baseline and the conclusion of the intervention (~10 weeks). Additionally, over weeks 8 and 9, participants will be invited for an in-person lab visit for a Trier Social Stress Test (TSST-OL) to assess reactivity to an acute social stressor.

This study aims to examine whether integrating mindfulness practice into a ten-week undergraduate-level biology course will enhance applied mindfulness and stress regulation capacity. We hypothesize that completing this ten-week course will (1) increase applied mindfulness, (2) increase self-efficacy in stress regulation, and (3) decrease perceived stress in response to an acute stressor.

Secondary analyses will also evaluate differential changes in individual well-being score components (including learning-related anxiety, self-compassion, social connectedness, alcohol use, media addiction, overall well-being, and physiological reactivity to an acute stressor).

Linear mixed effect models with a time and treatment interaction term and random intercepts by the participant will be fit to examine the first two hypotheses to account for repeated measurements and potential data missingness. To test the third hypothesis, we will compute the pre- to post-stress induction changes in subjective stress. Next, two-sample t-tests will be run on each change score to examine differences in responses to the stress challenge between the two groups. As sensitivity analyses, effect modification by baseline dispositional mindfulness, perceived stress over the last month, and severity of anxiety will be examined by including a three-way interaction term in the models to understand whether the intervention effect differs by these baseline characteristics. Further, the effect of the class on secondary outcomes will be explored with linear mixed-effect models. All analyses will consider a p-value < 0.05 as statistical significance.

ELIGIBILITY:
Inclusion criteria: 1. Undergraduate students who selected Biology 3: Mindful Physiology during the 2025 Spring term course enrollment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Applied Mindfulness | Baseline and intervention completion (~10 weeks)
  Students will complete the Applied Mindfulness Process Scale (AMPS) at baseline and post-intervention completion. The scale consists of 15 questions that quantify the application of mindfulness skills to navigate difficult situations and stressors in life. The AMPS encompasses three subscales: decentering, negative emotion regulation, and positive emotion regulation. The total scores are the sum across items. The total possible scores range from 0 to 60. Higher scores reflect a more active use of mindfulness practice in everyday life. The scale showed high internal validity with a Cronbach's α of 0.91 in 134 adults in the original study. Additionally, the application of mindfulness in stressful situations will be assessed during the Trier Social Stress Test (TSST) in our lab. Participants will report whether they have used mindfulness techniques during the stress challenge.
Stress Management Self-Efficacy | Baseline and intervention completion (~10 weeks)
  Participants will evaluate their confidence in managing stress with the Stress Management Self-Efficacy Scale (α = 0.86, N = 2292). The scale has four items, e.g., "I believe I have the ability to cope with the demands of my life." Additionally, students will answer three items from the Stress Management Self-Efficacy Measure on self-efficacy in recognizing the physiological responses to stress. The items are (1) I am confident identifying the causes of stress, (2) I am confident identifying physiological indicators of stress, and (3) I am confident predicting the consequences of stress. All items will be rated on a four-point Likert scale from 1 (strongly disagree) to 4 (strongly agree). A global score will be computed with the mean across the seven items (range: 1 to 4), with higher scores indicating greater self-efficacy in identifying and managing stress.
Perceived Stress in Response to an Acute Stressor | Intervention completion (~8 and 9 weeks)
  Stress reactivity will be assessed during an in-person lab visit with the online Trier Social Stress Test (TSST-OL). The TSST-OL is a computerized stress induction protocol, including 5 minutes of brief preparation, 5 minutes of public speaking (job interview), and 5 minutes of a math test in front of a panel of evaluators online. Our protocol will be modified to use a pre-recorded video of the panel of evaluators to give the impression of a live audience and minimize research assistant time while maintaining the conditions of the established TSST-OL. Perceived stress will be assessed at baseline (five minutes before the speech preparation) and immediately after the TSST with the Subjective Units of Distress Scale (SUDS). Participants will rate their level of distress from 0 (totally relaxed) to 100 (highest distress). Perceived stress reactivity will be operationalized as the difference between the post-TSST and baseline ratings.

SECONDARY OUTCOMES:
Self-Compassion | Baseline and intervention completion (~10 weeks)
  Self-compassion will be measured with the Self-Compassion Scale short-form (SCS-SF). This 12-item questionnaire evaluates how often one treats themselves with kindness rather than judgment during challenging moments. This instrument showed high internal validation in the original study (α ≥ .86) and correlated highly (r ≥ 0.97) with the original 33-item Self-Compassion Scale. The total possible score ranges from 1 to 5. Higher scores indicate more self-compassion.
Overall Well-Being | Baseline and intervention completion (~10 weeks)
  Overall well-being will be assessed with the ten-item Flourish measure. This self-report instrument has five domains: (1) life satisfaction (e.g., "In general, how happy or unhappy do you usually feel?"), (2) mental and physical health (e.g., "How would you rate your physical health?"), (3) meaning and purpose (e.g., "I understand my purpose in life."), (4) character and virtue (e.g., "I always act to promote good in all circumstances, even in difficult and challenging situations."), and (5) social relationships (e.g., "I am content with my friendships and relationships"). Items will be rated on a scale from 0 to 10, with higher scores reflecting more positive well-being. A total score will be computed by summing item responses (range: 0 to 50).
Social Connectedness | Baseline and intervention completion (~10 weeks)
  Social belongingness will be measured via the revised Social Connectedness Scale (SCS-r). Participants will rate 20 items on a six-point Likert scale from 1 (strongly disagree) to 6 (strongly agree), e.g., "I am able to relate to my peers." A total score will be computed by taking the sum across items. Possible scores range from 20 to 120, with 120 indicating the strongest sense of belongingness.
Mental Well-Being | Baseline and intervention completion (~10 weeks)
  Psychological well-being will be assessed with the 5-item World Health Organization Well-Being Index (WHO-5). Participants will rate five positively phrased items on subjective well-being, i.e., "I have felt cheerful and in good spirits." Responses are anchored from 0 (none of the time) to 5 (all the time). The total score is the sum of item responses ranging from 0 to 25, with 25 indicating the maximum possible mental well-being. The index has shown high internal consistency with α = 0.86 and test-retest reliability of r = 0.77 in 903 college students.
Resillience | Baseline and intervention completion (~10 weeks)
  Resilience to stress will be measured with the Brief Resilience Scale (BRS). The scale has six items on the ability to recover from difficulties in life, e.g., "I tend to bounce back quickly after hard times." Responses are anchored on a five-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The final score is the mean across the items, ranging from 1 to 5. Higher scores indicate more resilience. The scale demonstrated high internal validity with α ranging from 0.84 and 0.87 in two samples of US undergraduate students.
Learning-Related Anxiety | Baseline and intervention completion (~10 weeks)
  Anxiety around learning will be assessed with the learning-related anxiety subscale from the Achievement Emotions Questionnaire-Short Form (AEQ-S). Participants will rate four five-point Likert scales on feelings of anxiousness when studying, e.g., "I get tense and nervous while studying." The subscale showed adequate internal validity in the original study with an α of 0.72 in 180 adults (71% female, 58% White).
Social Media Addiction | Baseline and intervention completion (~10 weeks)
  Addictive use of social media will be examined with the Bergen Social Media Addiction Scale (BSMAS). Participants will rate six items reflecting elements of addiction to social media, e.g., "I spent a lot of time thinking about social media or planned use of social media (salience)" and "I felt an urge to use social media more and more (craving/tolerance)." Responses are anchored from 1 (very rarely) to 5 (very often). A total score will be computed by summing all item responses (range: 1 to 30). Higher scores indicate more addictive use of social media. The scale has shown adequate internal validity (α = 0.88, N = 23533 adults).
Alcohol Intake | Baseline and intervention completion (~10 weeks)
  Alcohol intake will be assessed via the Consumption subscale from the Alcohol Use Disorders Identification Test (AUDIT-C). The AUDIT-C has three items on the frequency and quantity of alcohol use. The total score is the sum across items, which range from 0 to 12, with higher scores indicating a higher risk of alcohol abuse or dependence. A score of 3 and above is indicative of possible risky drinking that warns of clinical concerns.
Physiological Stress in Response to an Acute Stressor | Intervention completion (~8 and 9 weeks)
  During the TSST, heart rate will be collected via a chest-worn monitor Polar H10 chest strap device (Polar Electro Oy, Kempele, Finland) and video-based photoplethysmography (PPG) (GoPro 9, San Mateo, US). The mean of the heart rate (HR), heart rate variability (HRV), and respiratory sinus arrhythmia (RSA) will be computed for three phases: the last 5 minutes of the baseline resting period, the last 3 minutes of the TSST, and the last 5 minutes of the recovery phase. Reactivity to the acute stressor will be operationalized as the differences in heart rate parameters during the TSST from the baseline. Recovery from the acute stressor will be operationalized as the difference between the recovery phase and baseline.

OTHER OUTCOMES:
Dispositional Mindfulness | Baseline and intervention completion (~10 weeks)
  Trait mindfulness will be assessed with the Five Facet Mindfulness Questionnaire (FFMQ), a 39-item questionnaire evaluating five distinct components of mindfulness: observation (8 items), description (8 items), aware actions (8 items), non-judging of inner experience (8 items), and non-reactivity to inner experience (7 items). The total score is the average across the five subscales. Possible scores range from 1 to 5, with higher scores indicating higher dispositional mindfulness.
Perceived Stress During the Last Month | Baseline and intervention completion (~10 weeks)
  Subjective stress in the last month will be measured with the ten-item Perceived Stress Scale (PSS-10). The scale evaluates individuals' perception of how uncontrollable and overloaded their lives have been in the past month, e.g., "In the past month, how often have you felt you were unable to control the important things in your life?" Participants will rate items on a five-point Likert scale from 0 (never) to 5 (very often). The possible scores range from 0 to 50; higher scores reflect more perceived stress. The scale has shown strong internal validity (α > 0.70) and test-retest reliability (r > 0.70) in a systematic review.
Anxiety | Baseline and intervention completion (~10 weeks)
  The severity of generalized anxiety disorder will be evaluated with the seven-item anxiety scale (GAD-7). The scale had high internal validity (α = 0.92) and test-retest reliability (interclass correlation = 0.83) in the original study. Item responses are anchored on a four-point Likert scale from 0 (not at all) to 3 (nearly every day). A total score will be computed by taking the sum of item responses. Possible scores range from 0 to 21, with higher scores reflecting more severe anxiety. A score of 8 and above indicates possible cases of GAD with a sensitivity of 83% and specificity of 84%.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Gilbert-Diamond, ScD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available to other researchers upon reasonable requests to the Principal Investigator with a data sharing agreement provided that the researchers have appropriate human subjects research approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available on October 1, 2026.
Access Criteria: Data Sharing Agreement Institutional Human Subjects Research Protocol Approval

REFERENCES:
- [Background] Heyers K, Pfeifer LS, Merz CJ, Stockhorst U, Gunturkun O, Wolf OT, Ocklenburg S. TSST-OL: Comparison between online and laboratory application and effects on empathy. Psychoneuroendocrinology. 2025 Jan;171:107211. doi: 10.1016/j.psyneuen.2024.107211. Epub 2024 Oct 11. PMID 39442231
- [Background] Schou Andreassen C, Billieux J, Griffiths MD, Kuss DJ, Demetrovics Z, Mazzoni E, Pallesen S. The relationship between addictive use of social media and video games and symptoms of psychiatric disorders: A large-scale cross-sectional study. Psychol Addict Behav. 2016 Mar;30(2):252-62. doi: 10.1037/adb0000160. PMID 26999354
- [Background] Stress and Quality of Life Among University Students: A Systematic Literature Review. Health Professions Education,
- [Background] US Preventive Services Task Force; Curry SJ, Krist AH, Owens DK, Barry MJ, Caughey AB, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Kubik M, Landefeld CS, Mangione CM, Silverstein M, Simon MA, Tseng CW, Wong JB. Screening and Behavioral Counseling Interventions to Reduce Unhealthy Alcohol Use in Adolescents and Adults: US Preventive Services Task Force Recommendation Statement. JAMA. 2018 Nov 13;320(18):1899-1909. doi: 10.1001/jama.2018.16789. PMID 30422199
- [Background] VanderWeele TJ. On the promotion of human flourishing. Proc Natl Acad Sci U S A. 2017 Aug 1;114(31):8148-8156. doi: 10.1073/pnas.1702996114. Epub 2017 Jul 13. PMID 28705870
- [Background] Zhang Z, Luu BCP, Gilbert-Diamond D. Acceptability, engagement, and preliminary efficacy of a college human physiology course with integrated mindfulness practice to support student wellbeing. Front Psychol. 2024 Aug 14;15:1365778. doi: 10.3389/fpsyg.2024.1365778. eCollection 2024. PMID 39205975
- [Background] Wunsch K, Fiedler J, Bachert P, Woll A. The Tridirectional Relationship among Physical Activity, Stress, and Academic Performance in University Students: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jan 16;18(2):739. doi: 10.3390/ijerph18020739. PMID 33467118
- [Background] Sawatzky RG, Ratner PA, Richardson CG, Washburn C, Sudmant W, Mirwaldt P. Stress and depression in students: the mediating role of stress management self-efficacy. Nurs Res. 2012 Jan-Feb;61(1):13-21. doi: 10.1097/NNR.0b013e31823b1440. PMID 22166906
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Plummer F, Manea L, Trepel D, McMillan D. Screening for anxiety disorders with the GAD-7 and GAD-2: a systematic review and diagnostic metaanalysis. Gen Hosp Psychiatry. 2016 Mar-Apr;39:24-31. doi: 10.1016/j.genhosppsych.2015.11.005. Epub 2015 Nov 18. PMID 26719105
- [Background] Pirzada P, Wilde A, Doherty GH, Harris-Birtill D. Ethics and acceptance of smart homes for older adults. Inform Health Soc Care. 2022 Jan 2;47(1):10-37. doi: 10.1080/17538157.2021.1923500. Epub 2021 Jul 9. PMID 34240661
- [Background] Nyklicek I, Mommersteeg PM, Van Beugen S, Ramakers C, Van Boxtel GJ. Mindfulness-based stress reduction and physiological activity during acute stress: a randomized controlled trial. Health Psychol. 2013 Oct;32(10):1110-3. doi: 10.1037/a0032200. Epub 2013 Mar 25. PMID 23527521
- [Background] Johnson BT, Acabchuk RL, George EA, Nardi W, Sun S, Salmoirago-Blotcher E, Scharf J, Loucks EB. Mental and Physical Health Impacts of Mindfulness Training for College Undergraduates: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Mindfulness (N Y). 2023 Sep;14(9):2077-2096. doi: 10.1007/s12671-023-02212-6. Epub 2023 Sep 22. PMID 38250521
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Galante J, Dufour G, Vainre M, Wagner AP, Stochl J, Benton A, Lathia N, Howarth E, Jones PB. A mindfulness-based intervention to increase resilience to stress in university students (the Mindful Student Study): a pragmatic randomised controlled trial. Lancet Public Health. 2018 Feb;3(2):e72-e81. doi: 10.1016/S2468-2667(17)30231-1. Epub 2017 Dec 19. PMID 29422189
- [Background] Dawson AF, Brown WW, Anderson J, Datta B, Donald JN, Hong K, Allan S, Mole TB, Jones PB, Galante J. Mindfulness-Based Interventions for University Students: A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Appl Psychol Health Well Being. 2020 Jul;12(2):384-410. doi: 10.1111/aphw.12188. Epub 2019 Nov 19. PMID 31743957
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717